CLINICAL TRIAL: NCT00078663
Title: The Effect of a Systemic Oral Care Program on Reducing Exposure to Oropharyngeal Pathogens in Critically III Patients
Brief Title: Oral Care to Reduce Mouth and Throat Infections in Critically Ill Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040130; 04-CC-0130
Record Dates: First submitted 2004-03-03; First posted 2004-03-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-08-16

CONDITIONS: Critical Illness
Keywords: Oral Care; ICU; Pneumonia; Pathogens; Intubation; Intubated; Oral Hygiene; Intensive Care
MeSH Terms: conditions — Critical Illness; Pneumonia | interventions — Dental Care Team

INTERVENTIONS:
Behavioral: Oral Care

SUMMARY:
This study will evaluate whether a program of systematic oral care can help prevent hospital-acquired respiratory infections in patients in intensive care units. Such infections occur five times more often in critically ill patients compared with patients in general hospital wards and result in longer hospital stays and an increased risk of death. The rate of respiratory infection among critically ill patients correlates strongly with the presence of disease-causing bacteria in the mucosal areas of the mouth, gums, and teeth, indicating that assiduous oral care is especially important in this patient population. This study will compare a program of meticulous oral care using oral assessments taught by a dentist and dental hygienist with the standard care typically given in intensive care units.

Critically ill patients 18 years of age and older who are hospitalized in an intensive care unit for 3 or more days and whose oral hygiene is dependent on hospital care providers may be eligible for this study. Patients will be recruited from intensive care units at four Washington, D.C., area hospitals - Suburban Hospital, Washington Hospital Center, Inova Fairfax Hospital, and Winchester Medical Center.

Participants will have their lips, mouth, gums, teeth, and saliva examined several times a day to determine their optimum oral care. They will receive standard care, such as flossing, brushing, rinsing with a mouthwash, and possibly use of an antiseptic spray that prevents bacteria from clinging to the teeth. Small samples of saliva (less than one-fourth of a teaspoon) and dental plaque will be collected the day the patient is admitted to the intensive care unit and again on days 3 and 5 of their stay in the unit. The saliva sample is collected with a small suction tube placed in the corner of the mouth; the plaque specimen is collected by gliding a tiny piece of paper over the surface of a front tooth. The samples will be examined for any bacteria not normally found in saliva.

DETAILED DESCRIPTION:
Critically ill patients, especially those that require endotracheal intubation, have the greatest risk of any hospitalized patient for acquiring nosocomial pneumonia. Nosocomial pneumonia, in this population, produces a substantial increase of mortality and morbidity. The literature suggests the causative pathway is aspiration of oropharyngeal pathogens found in dental plaque. The build-up of dental plaque has been significantly associated with subsequent nosocomial respiratory infections. Thus, prevention of pathogens colonization in the oropharyngeal cavity could be an effective infection control measure.

Dental plaque once it reaches a critical thickness, acts as a reservoir for both aerobic and anaerobic pathogens. Failure to remove plaque begins a complex cascade of biological activity by which pathogens adhere to mucosal and tooth surfaces and pathogen overgrowth ensues. Additionally, neglected or insufficient mouth care is the foremost predisposing factor to oral conditions such as gingivitis, mucositis, and stomatitis which supply additional ports of entry for pathogens.

There are only a handful of studies that compare the frequency and type of oral hygiene required to prevent or decrease oropharyngeal colonization. A recent pilot study, 01-CC-0207, compared oral care provision in two intensive care units (ICU) in the Clinical Center. The test ICU offered meticulous oral hygiene through a system of regular oral assessments taught by a dentist and dental hygienist. The score from the assessment determined the type and frequency of oral care. The control ICU gave standard care typical of the ICU community. Plaque and saliva assays were collected from the enrolled patients. Significantly lower Beck scores and lower colony forming organisms in the specimens was achieved in the test ICU on day 3, p less than 0.03 and p less than 0.001 respectively.

This protocol will expand the pilot into a prospective randomized assigned trial conducted at four hospitals in the Washington D.C. area. These hospitals have ICUs more representative of ICU's nation-wide. This study will test the effectiveness of a comprehensive and systematic oral care program to reduce the oral assessment scores, mucosal plaque scores, and the amount of pathogen inoculum present in the saliva and plaque. Intubated and non-intubated patients will be compared as well as meticulous care with or without the addition of the oral antiseptic, chlorhexidine. Consistency of practice performance will also be evaluated when nursing staff has dentist/hygienist instruction and monitoring versus the traditional nurse instruction.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male or female adult ICU patients whose oral hygiene is dependent upon hospital care providers.
* Expected length of ICU stay is greater than or equal to 3 days.
* Any gender and ethnicity.

EXCLUSION CRITERIA:

* Individuals and or responsible family members who are unable to provide consent.
* Any individual under the age of 18 years.
* Any individual whose expected admission is less than 3 days.
* Adult ICU patients whose admission CPIS score is greater than 6.
* Individuals who are able to provide own oral care.
* Individuals who have oral surgery that requires specialized oral care and assessment.
* Edentulous patients.
* Any patient with a prosthetic heart valve or who routinely takes prophylactic antibiotics before routine dental procedures.
* Any patient with a known allergy to chlorhexidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2004-03-02; Primary Completion 2007-12-28 (Actual); Study Completion 2011-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Inova Fairfax Hospital, Fairfax, Virginia
  - Winchester Medical Center, Winchester, Virginia

REFERENCES:
- [Background] Collard HR, Saint S, Matthay MA. Prevention of ventilator-associated pneumonia: an evidence-based systematic review. Ann Intern Med. 2003 Mar 18;138(6):494-501. doi: 10.7326/0003-4819-138-6-200303180-00015. PMID 12639084
- [Background] Valles J, Mesalles E, Mariscal D, del Mar Fernandez M, Pena R, Jimenez JL, Rello J. A 7-year study of severe hospital-acquired pneumonia requiring ICU admission. Intensive Care Med. 2003 Nov;29(11):1981-8. doi: 10.1007/s00134-003-2008-4. Epub 2003 Sep 10. PMID 13680109
- [Background] Eggimann P, Hugonnet S, Sax H, Touveneau S, Chevrolet JC, Pittet D. Ventilator-associated pneumonia: caveats for benchmarking. Intensive Care Med. 2003 Nov;29(11):2086-9. doi: 10.1007/s00134-003-1991-9. Epub 2003 Sep 3. PMID 12955177